CLINICAL TRIAL: NCT03377036
Title: Prospective Randomized Comparison of Digital Breast Tomosynthesis Plus Synthesized Images Versus Standard Full-field Digital Mammography in Population-based Screening (TOSYMA)
Brief Title: Breast Cancer Screening: Digital Breast Tomosynthesis Versus Digital 2D Mammography
Acronym: TOSYMA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: UKM14_0016; HE1646/5-1 and HE1646/5-2 (Other Grant/Funding Number: German Research Foundation (DFG))
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Screening
Keywords: Breast Cancer; Population-based Screening; Digital Breast Tomosynthesis plus synthesized Mammography; Reconstructed Mammography; Full-Field Digital Mammography (FFDM); Multicentric Randomized Controlled Trial; Diagnostic Performance; Recall Rate; Interval Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either Digital Breast Tomosynthesis plus synthesized 2D mammograms (DBT+s2D) or 2D Full-Field Digital Mammography (2D-FFDM)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBT+s2D (Experimental): Digital breast tomosynthesis plus synthesized 2D mammograms
  Interventions: Diagnostic Test: DBT+s2D
- 2D-FFDM (Active Comparator): 2D full-field digital mammography
  Interventions: Diagnostic Test: 2D-FFDM

INTERVENTIONS:
Diagnostic Test: DBT+s2D — Digital breast tomosynthesis plus synthesized 2D mammograms
  Arms: DBT+s2D
Diagnostic Test: 2D-FFDM — 2D full-field digital mammography
  Arms: 2D-FFDM

SUMMARY:
This study is a randomized, multicenter, multivendor, controlled, diagnostic superiority trial to compare digital breast tomosynthesis plus synthesized 2D mammograms (DBT+s2D) versus standard 2D full-field digital mammography (2D-FFDM) regarding the effectiveness as screening modality.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate whether digital breast tomosynthesis plus synthesized 2D mammograms leads to a relevant increase in the detection rate of screening-detected invasive cancers compared to 2D full-field digital mammography in routine screening according to the European Guidelines. Furthermore, the incidence rate of interval cancers within a 24 months interval after screening will be compared between both study arms in order to investigate the potential for overdiagnosis.

According to the pre-defined order of both primary endpoints and the primary objective of the study in the planning phase, the initial sample size calculation was based solely on the first primary endpoint (invasive breast cancer detection rate). Given the increasing national and international attention of interval cancers to assess the impact of potential overdiagnosis caused by tomosynthesis, we have planned a sample size increase from 80,000 to 120,000 study participants to achieve a reasonable statistical power for the evaluation of both primary endpoints. The revised sample size calculation was carried out without knowledge of the data from the currently recruiting TOSYMA study, i.e. all planning assumptions were based on external data that do not belong to the ongoing study.

ELIGIBILITY:
Inclusion Criteria:

* Women eligible to participate in the National Mammography Screening Program of Germany
* Informed decision for mammography screening
* Written informed consent
* No prior participation in the TOSYMA trial

Exclusion Criteria:

* Breast cancer up to 5 years prior to study invitation
* Previous mammography examination < 12 months,
* Breast implants

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 99689 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Detection rate of invasive breast cancers | Routine screening visit
  Number of women with screening-detected invasive breast cancer divided by the number of all women screened. A screening-detected breast cancer is classified as invasive carcinoma if the pT category (pathological tumor size) of the TNM classification falls into one of the following categories: pT1mic, pT1a, pT1b, pT1c, pT1, pT2, pT3, pT4a, pT4b, pT4c, pT4d, pT4, pTX (for evaluation purpose pTX defines histologically approved invasive breast cancer with missing tumor diameter) or the final pathological categorization has been done after neoadjuvant therapy (ypT), implying an invasive cancer prior to therapy.
Cumulative 24 months incidence of interval cancers | 24 months after routine screening visit
  The 24 months incidence of interval cancers is defined as the number of women that develop a ductal carcinoma in situ or an invasive breast cancer in the 24 months interval after a negative screening examination divided by the number of all women with a negative screening result.

SECONDARY OUTCOMES:
Detection rate of ductal carcinoma in situ (DCIS) | Routine screening visit
  Number of women with screening-detected ductal carcinoma in situ (if the pT category of the TNM classification falls into the category pTis) divided by the number of all women screened.
Detection rate of tumor category pT1 | Routine screening visit
  Number of women with screening-detected invasive breast cancers of the category pT1 divided by the number of all women screened. A screening-detected breast cancer is classified as breast cancer of tumor category pT1 if tumor size is ≤ 20 mm in greatest dimension and the respective pT subcategory of the pTNM classification is one of the following: pT1mic, pT1a, pT1b, pT1c, pT1.
Recall rate for further assessment | Routine Screening Visit
  Number of women with recalls for further assessment divided by the number of all women screened.
Positive predictive value of recall for further assessment (PPV1) | Routine screening visit
  Number of women with screening-detected malignancies (ductal carcinoma in situ or invasive breast cancer) divided by the number of women with recalls for further assessment.
Cumulative 12 months incidence of interval cancers | 12 months after routine screening visit
  The 12 months incidence of interval cancers is defined as the number of women that develop a ductal carcinoma in situ or an invasive breast cancer in the 12 months interval after a negative screening examination divided by the number of all women with a negative screening result.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Heindel, MD, PhD, Principal Investigator — University Clinic for Radiology, University of Muenster / University Hospital Muenster
Locations (21):
- Germany (21):
  - Screening-Einheit Hannover; Mammographie-Einheit Hannover, Hanover, Lower Saxony
  - Screening-Einheit Niedersachsen Nordost; Mammographie-Einheit Lüneburg, Lüneburg, Lower Saxony
  - Screening-Einheit Niedersachsen Nord; Mammographie-Einheit Stade, Stade, Lower Saxony
  - Screening-Einheit Niedersachsen Mitte; Mammographie-Einheit Vechta, Vechta, Lower Saxony
  - Screening-Einheit Niedersachsen Nordwest; Mammographie-Einheit Wilhelmshaven, Wilhelmshaven, Lower Saxony
  - Screening-Einheit Aachen-Düren-Heinsberg; Mammographie-Einheit Aachen, Aachen, North Rhine-Westphalia
  - Referenz-Screening-Einheit Münster-Nord/Warendorf; Mammographie-Einheit Ahlen, Ahlen, North Rhine-Westphalia
  - Screening-Einheit Köln rechtsrheinisch, Leverkusen, Rhein.-Berg. Kreis, Oberbergischer Kreis; Mammographie-Einheit Bergisch Gladbach, Bergisch Gladbach, North Rhine-Westphalia
  - Screening-Einheit Bielefeld, Gütersloh; Mammographie-Einheit Bielefeld, Bielefeld, North Rhine-Westphalia
  - Screening-Einheit Münster-Süd; Mammographie-Einheit Coesfeld, Coesfeld, North Rhine-Westphalia
  - Screening-Einheit Duisburg; Mammographie-Einheit Duisburg, Duisburg, North Rhine-Westphalia
  - Screening-Einheit Gelsenkirchen, Kreis Recklinghausen, Bottrop; Mammographie-Einheit Gelsenkirchen, Gelsenkirchen, North Rhine-Westphalia
  - Screening-Einheit Minden-Lübbecke, Herford; Mammographie-Einheit Herford, Herford, North Rhine-Westphalia
  - Screening-Einheit Mönchengladbach, Krefeld, Viersen; Mammographie-Einheit Krefeld, Krefeld, North Rhine-Westphalia
  - Screening-Einheit Höxter, Paderborn, Soest; Mammographie-Einheit Lippstadt, Lippstadt, North Rhine-Westphalia
  - Referenz-Screeening-Einheit Münster-Nord/Warendorf; Mammographie-Einheit Münster-Nord, Münster, North Rhine-Westphalia
  - Screening-Einheit Münster-Süd; Mammographie-Einheit Münster, Münster, North Rhine-Westphalia
  - Screening-Einheit Höxter, Paderborn, Soest; Mammographie-Einheit Paderborn, Paderborn, North Rhine-Westphalia
  - Screening-Einheit Märkischer Kreis, Hamm, Unna; Mammographie-Einheit Schwerte, Schwerte, North Rhine-Westphalia
  - Screening-Einheit Raum Bergisch Land/Kreis Mettmann; Mammographie-Einheit Solingen-Mitte, Solingen, North Rhine-Westphalia
  - Screening-Einheit Raum Bergisch Land/Kreis Mettmann; Mammographie-Einheit Wuppertal-Elberfeld, Wuppertal, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weigel S, Gerss J, Hense HW, Krischke M, Sommer A, Czwoydzinski J, Lenzen H, Kerschke L, Spieker K, Dickmaenken S, Baier S, Urban M, Hecht G, Heidinger O, Kieschke J, Heindel W. Digital breast tomosynthesis plus synthesised images versus standard full-field digital mammography in population-based screening (TOSYMA): protocol of a randomised controlled trial. BMJ Open. 2018 May 14;8(5):e020475. doi: 10.1136/bmjopen-2017-020475. PMID 29764880
- [Derived] Weigel S, Heindel W, Hense HW, Decker T, Gerss J, Kerschke L; TOSYMA Screening Trial Study Group. Breast Density and Breast Cancer Screening with Digital Breast Tomosynthesis: A TOSYMA Trial Subanalysis. Radiology. 2023 Feb;306(2):e221006. doi: 10.1148/radiol.221006. Epub 2022 Oct 4. PMID 36194110
- [Derived] Heindel W, Weigel S, Gerss J, Hense HW, Sommer A, Krischke M, Kerschke L; TOSYMA Screening Trial Study Group. Digital breast tomosynthesis plus synthesised mammography versus digital screening mammography for the detection of invasive breast cancer (TOSYMA): a multicentre, open-label, randomised, controlled, superiority trial. Lancet Oncol. 2022 May;23(5):601-611. doi: 10.1016/S1470-2045(22)00194-2. Epub 2022 Apr 12. PMID 35427470
- See also: BMJ Open — http://bmjopen.bmj.com/content/8/5/e020475